CLINICAL TRIAL: NCT02158247
Title: Determining the Depth of Endotracheal Tube Insertion
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Saecheol Oh, Associate Professor, The Catholic University of Korea
Other Study IDs: DJSMAN-01
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Endotracheal Intubation; Individualized Depth of Endotracheal Intubation

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Conventional group, Touch and Read group

SUMMARY:
1. Airway length from the medial incisor to carina is divided into four segments ; the length from medial incisor to mouth angle, mouth angle to epiglottis, epiglottis to vocal cords and vocal cords to carina.
2. Determining the mean length of each segments with the direct laryngoscope, videolaryngoscope and fiberoptic bronchoscope at the time of endotracheal intubation.
3. Making a new formula to determine the proper individualized depth of intubation on the basis of the length of segments
4. Virtual experiment : comparing the new formula with conventional method of determining the depth of endotracheal intubation

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to take general anesthesia with endotracheal intubation

Exclusion Criteria:

* Patients undergoing general anesthesia with face mask ventilation or laryngeal mask airway

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are taking operation in the university hospital
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and Pain Medicine, Daejeon St Mary's hospital, Daejeon, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Tough and Read Group: This is a virtual experiment based on the anthropometry of the airway length. Conventional group : We defined the conventional group as patients who are intubated on the depth of 25cm for male and 23 cm fo female from the medial incisor virtually.
  Touch and read group : Depth of intubation was determined on the measurement of the airway length of each patient. In touch and read group, the depth of intubation was determined by the sum of the length from the mouth angle to epiglottis tip, the length from the epiglottis tip to vocal cords and 8cm for the endotracheal tube #7.0. Length from the mouth angle to epiglottis tip is determined at the time of intubation with specially scaled endotracheal tube.
Period: Overall Study
Arm/Group | Tough and Read Group
Started | 181
Completed | 176
Not Completed | 5
Not completed — Invisible vocal cords | 5

BASELINE CHARACTERISTICS:
Population: Male : 69, Female : 107
Groups:
- Touch and Read Group(Male): This is a virtual experiment based on the anthropometry of the airway length. We defined the conventional group as patients who are intubated on the depth of 25cm for male and 23 cm fo female from the medial incisor virtually.
  Touch and read group : Depth of intubation was determined on the measurement of the airway length of each patient. In touch and read group, the depth of intubation was determined by the sum of the length from the mouth angle to epiglottis tip, the length from the epiglottis tip to vocal cords and 8cm for the endotracheal tube #7.0. Length from the mouth angle to epiglottis tip is determined at the time of intubation with specially scaled endotracheal tube.
- Touch and Read Group(Female): female
- Total: Total of all reporting groups
Arm/Group | Touch and Read Group(Male) | Touch and Read Group(Female) | Total
Number analyzed (Participants) | 69 | 107 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 82 | 144
  >=65 years | 7 | 25 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 107 | 107
  Male | 69 | 0 | 69

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Airway Length Between Male and Female
Description: Airway length is defined the distance from medial incisor to carina. It is divided into four parts. It is medial incisor to mouth angle, mouth angle to epiglottis tip, epiglottis tip to vocal cords and vocal cords to carina.
Time Frame: Endotracheal intubation time
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Airway Length for Male | Airway Length of Female
Number analyzed (Participants) | 69 | 107
Centimeters
  Medial incisor to mouth angle | 0.9 (0.5) | 1.1 (0.5)
  Mouth angle to epiglottis tip | 9.1 (1.0) | 8.3 (1.0)
  Epiglottis tip to vocal cords | 4.4 (0.9) | 3.6 (0.9)
  Vocal cords to carina | 11.9 (1.3) | 11.2 (1.2)
  Medial incisor to carina | 26.4 (1.9) | 24.2 (1.5)

2. Secondary Outcome: Comparison Between Conventional Method and Touch and Read Method for Risk Group of Male
Description: Normal group is defined as the patients whose airway length from medial incisor to carina is below 25cm.
  Conventional method : depth of intubation is 23cm at the medial incisor for male.
  Touch and read method : depth of intubation is calculated as follow : length from mouth angle to epiglottis tip plus 12.5cm for male.
Time Frame: Endotracheal intubation time
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Conventional Method for Risk Group of Male | Touch and Read for Risk Group of Male
Number analyzed (Participants) | 15 | 15
Centimeters
  Tube tip to carina | 0.7 (1.4) | 2.0 (1.2)
  Vocal cords to cuff | 3.5 (1.4) | 2.3 (1.1)

3. Secondary Outcome: Comparison Between Conventional Method and Touch and Read Method for Normal Group of Male
Description: Normal group is defined as the patients whose airway length from medial incisor to carina is over 25cm.
  Conventional method : depth of intubation is 23cm at the medial incisor for male.
  Touch and read method : depth of intubation is calculated as follow : length from mouth angle to epiglottis tip plus 12.5cm for male.
Time Frame: Endotracheal intubation time
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Conventional Method for Normal Group of Male | Touch and Read for Normal Group of Male
Number analyzed (Participants) | 54 | 54
Centimeters
  Tube tip to carina | 4.1 (1.2) | 4.4 (1.2)
  Vocal cords to cuff | 2.3 (0.8) | 2.0 (1.0)

4. Secondary Outcome: Comparison Between Conventional Method and Touch and Read Method for Risk Group of Female
Description: Risk group is defined as the patients whose airway length from medial incisor to carina is below 23cm.
  Conventional method : depth of intubation is 21cm at the medial incisor for female.
  Touch and read method : depth of intubation is calculated as follow : length from mouth angle to epiglottis tip plus 11.5cm for female.
Time Frame: Endotracheal intubation time
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Conventional Method for Risk Group of Female | Touch and Read for Risk Group of Female
Number analyzed (Participants) | 24 | 24
Centimeters
  Tube tip to carina | 1.2 (1.0) | 1.9 (1.1)
  Vocal cords to cuff | 2.7 (0.9) | 2.0 (0.9)

5. Secondary Outcome: Comparison Between Conventional Method and Touch and Read Method for Normal Group of Female
Description: Normal group is defined as the patients whose airway length from medial incisor to carina is over 23cm.
  Conventional method : depth of intubation is 21cm at the medial incisor for female.
  Touch and read method : depth of intubation is calculated as follow : length from mouth angle to epiglottis tip plus 11.5cm for female.
Time Frame: Endotracheal intubation time
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Conventional Method for Normal Group of Female | Touch and Read for Normal Group of Female
Number analyzed (Participants) | 83 | 83
Centimeters
  Tube tip to carina | 3.8 (1.0) | 3.8 (1.0)
  Vocal cords to cuff | 1.8 (0.9) | 1.9 (1.0)

6. Primary Outcome: Airway Length vs Height in Male
Time Frame: Endotracheal intubation time
Measure: Mean (Standard Deviation); unit: Centimeters
Groups:
- Airway Length vs Height in Male: Relationship between airway length and their height are analyzed with linear regression.
  Airway length is defined the distance from mouth angle to carina. Additionally it is divided into three parts, from mouth angle to epiglottis tip, epiglottis tip to vocal cords and vocal cords to carina.
Arm/Group | Airway Length vs Height in Male
Number analyzed (Participants) | 69
Centimeters
  Mouth angle to carina | 25.5 (1.8)
  Mouth angle to epiglottis tip | 9.1 (1.0)
  Epiglottis tip to vocal cords | 4.4 (0.9)
  Vocal cords to carina | 11.9 (1.3)
  Male height | 168 (7.4)

7. Primary Outcome: Airway Length vs Height in Female
Time Frame: Endotracheal intubation time
Measure: Mean (Standard Deviation); unit: Centimeters
Groups:
- Female Airway Length vs Height: Relationship between airway length and their height are analyzed with linear regression.
  Airway length is defined the distance from mouth angle to carina. Additionally it is divided into three parts, from mouth angle to epiglottis tip, epiglottis tip to vocal cords and vocal cords to carina.
Arm/Group | Female Airway Length vs Height
Number analyzed (Participants) | 107
Centimeters
  Mouth angle to carina | 23.2 (1.5)
  Mouth angle to epiglottis tip | 8.3 (1.0)
  Epglottis tip to vocal cords | 3.6 (0.9)
  Vocal cords to carina | 11.2 (1.2)
  Female height | 156.4 (5.2)

ADVERSE EVENTS:
Arm/Group | Touch and Read Group(Male) | Touch and Read Group(Female)
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/110
Other Adverse Events (participants affected / at risk) | 0/71 | 0/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Touch and Read Group(Male) (N=71) | Touch and Read Group(Female) (N=110)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Adverse events were not collected for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No